CLINICAL TRIAL: NCT05271747
Title: Prospective Study to Determine the Factors Influencing Infant Colic Course in Infants Taking Probiotics
Brief Title: Prospective Study to Determine the Factors Influencing Infant Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AB Biotics, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro-care 2
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2024-03

CONDITIONS: Infant Colic
Keywords: Infant colic, probiotic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: Randomized, multicentric, single-blind trial in infants between 2 and 12 weeks of age diagnosed with infant colic, who will be allocated to receive one of the two comercialized probiotic products B. Longum and P. Pentosaceus (branch one) or L. Reuteri (branch two) for 21 days
Who Masked: Investigator
Masking Description: Both probiotic products will be provided in their commercial form. Both products will be individually placed inside opaque bags so that the investigator can not recognize the external case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AB- Kolicare (Active Comparator): Probiotic multi-strain formulation comprising Bifidobacterium longum CECT7894 and Pediococcus pentosaceus CECT8330 in sunflower oil. Probiotic strains have Qualified Presumption of Safety (QPS) status by European Food Safety Authority
  Interventions: Dietary Supplement: AB-Kolicare
- Reuteri gotas (Active Comparator): Probiotic single-strain formulation comprising Lactobacillus reuteri DSM17938 in sunflower oil and medium-chain triglyceride oil. Probiotic strains have Qualified Presumption of Safety (QPS) status by European Food Safety Authority
  Interventions: Dietary Supplement: Reuteri gotas

INTERVENTIONS:
Dietary Supplement: AB-Kolicare — Probiotic multi-strain formulation containing Bifidobacterium longum CECT7894 and Pediococcus pentosaceus CECT8830 for 21 days, 5 drops/day preferably during the first intake of milk
  Arms: AB- Kolicare
Dietary Supplement: Reuteri gotas — Probiotic single-strain formulation containing Lactobacillus reuteri DSM17938 for 21 days, 5 drops/day before or after any daily meal.
  Arms: Reuteri gotas

SUMMARY:
Randomized study to determine the effect of a commercialized combination of 2 probiotic strains (Bifidobacterium Longum and Pediococcus pentosaceus) and the impact of feeding type in babies diagnosed with colic under Roma IV criteria when administered for 21 days.

DETAILED DESCRIPTION:
Randomized, single-blind, interventional study with two parallel groups to determine the effect of two different commercialized probiotic products (Lactobacillus reuteri or a combination of two different strains (Bifidobacterium longum and Pediococcus pentosaceus)) and the impact of feeding type in babies diagnosed with colic under Roma IV criteria. Infants meeting selection criteria are randomized 1:1 and stratified according to the type of feeding (breastfed or formula).

Probiotics are administered once a day (5 drops) for 21 days. Parents must document clinical parameters during this 21 days. This parameters include colic-related symptoms, other functional gastrointestinal disorders symptoms, parental anxiety and adverse events.

Moreoever, stool samples are collected to determine intestinal microbiota and calprotectin levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants from 2 to 12 weeks of age
* Infants diagnosed with infant colic following Roma IV criteria for clinical research
* Gestational age greater or equal to 37 weeks
* Birth weight greater than 2100 g
* Exclusively breastfed or formula fed with a maximum of one daily intake of breast milk.

Exclusion Criteria:

* Infants that are fed with solid food.
* Infants whose parents can not appropriately follow the requirements of the study.
* Antibiotics or probiotics administration to the infant (including infant formula with probiotics) 2 weeks prior the inclusion in the study.
* Breastfed infants whose mothers have taken antibiotics and/or probiotics 2 weeks prior the inclusion in the study.
* Infants fed extensively hydrolyzed infant formula
* Specific medication use for the treatment of functional digestive disorder: antacids (IBP type or H2 blockers), laxative Polyethylene glycol (8PEG), lactulose, magnesia), lactase or simeticone.
* Infants going through therapies related with acupuncture, homeopathy, medicinal herbs, or taking anti-inflammatory or antispasmodic drugs.

Ages: 2 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 112 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Duration of crying and fussing | 21 days
  Change on daily crying and fussing minutes measured through Barr ( Barr et al., 1988).validated crying and fussing scale. The Barr scale consists of a 24 hours dairy where parents paint number of hours crying and fussing every day. Results show the number of hours of crying and fussing per day.
Percent of responders | 7, 14, 21 days
  Percent of subjects whose change in crying time is equal or larger than 50% from baseline

SECONDARY OUTCOMES:
Number of regurgitations | 21 days
  Change in daily number of regurgitations
Bowel movements | 21 days
  Change in daily number of bowel movements
Food intake | 21 days
  Frequency of food intake
Parent's anxiety and depression | baseline, day 21
  Change in parent's anxiety and depression score measured through Hospital Anxiety and Depression Scale (HADS). The HADS questionnaire has 7 items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Fecal microbiome | baseline, day 21
  Changes on fecal microbiome evaluated by RNA ribosomal 16S genes analysis
Fecal calprotectin | baseline, day 21
  Change on calprotectin in feces
Adverse events | 21 days
  Frequency of adverse events reported on dairy report form after randomization and until day 21

CONTACTS AND LOCATIONS:
Locations (4):
- Hospital Medica Sur, room 108, tower 2, Mexico City, Mexico
- Spain (3):
  - University Hospital Santa Lucía, Cartagena, Murcia
  - HM Hospitals, Barcelona
  - Hm Hospitals, Madrid

REFERENCES:
- [Background] Drossman DA, Hasler WL. Rome IV-Functional GI Disorders: Disorders of Gut-Brain Interaction. Gastroenterology. 2016 May;150(6):1257-61. doi: 10.1053/j.gastro.2016.03.035. No abstract available. PMID 27147121
- [Derived] Moreno-Villares JM, Andrade-Platas D, Soria-Lopez M, Colome-Rivero G, Catalan Lamban A, Martinez-Figueroa MG, Espadaler-Mazo J, Valverde-Molina J. Comparative efficacy of probiotic mixture Bifidobacterium longum KABP042 plus Pediococcus pentosaceus KABP041 vs. Limosilactobacillus reuteri DSM17938 in the management of infant colic: a randomized clinical trial. Eur J Pediatr. 2024 Dec;183(12):5371-5381. doi: 10.1007/s00431-024-05806-x. Epub 2024 Oct 11. PMID 39390276